CLINICAL TRIAL: NCT05432817
Title: PTSD Treatment for Incarcerated Men and Women: WPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-0630: WPP; A538900 (Other: UW Madison); Protocol Version 5/21/2025 (Other: UW Madison)
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: PTSD
Keywords: Group therapy; Incarcerated Individuals
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two therapy-intervention groups: CPT or active waitlit control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy (CPT) group (Experimental): Participant groups to receive CPT to treat PTSD
  Interventions: Behavioral: Cognitive Processing Therapy
- Waitlist Control (No Intervention): Participant groups will provide data as a control group first, and will then receive CPT to treat PTSD

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT: a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered over 12 sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes homework assignments. For this study, CPT will be conducted in groups.
  Arms: Cognitive Processing Therapy (CPT) group

SUMMARY:
Study examining the psychological response to group Cognitive Processing Therapy (CPT) in incarcerated men and women with Post-traumatic stress disorder (PTSD). The study will be conducted in male and female incarcerated populations and will include 2 groups of individuals for both CPT and waitlist control in both populations (180 participants total).

DETAILED DESCRIPTION:
Overall Study Objectives:

The primary objectives of this project include:

1. Determine the effectiveness of CPT in reducing PTSD symptom severity;
2. Identify putative psychological mechanisms of response to CPT through pre-, mid-, and post-intervention measures of PTSD symptom severity as well as measures of hopelessness, self-blame, and negative self-related thoughts.

Prior to beginning any study procedures, informed consent will be obtained orally and in writing. During the informed consent process, eligible participants will be provided with detailed information about the study, including their right to refuse or discontinue participation at any time and the fact that their decision to participate or decline will have no bearing on their standing within the criminal justice system.

Potential participants will be contacted by calling them over the phone system within the prison. When they arrive to the private testing room, they are asked if they would like to learn about the study and potentially participate. If so, participants undergo consent.

Eligible participants will complete the PCL-5 to ascertain current PTSD symptomology and probable diagnosis. This assessment will take approximately 90 minutes.

Participants will be randomly assigned to the CPT or the active control groups. The CPT group will engage in 10 to 12, 90-minute treatment sessions (up to 18 hours total). With the optional opportunity to take 15-20 minutes after each session to de-stress and calm down if necessary. These sessions will take place over 6 to 12 weeks, depending on session frequency. CPT group-members are also asked to complete weekly homework (approximately 12 hours total). A maximum of 10 participants, but no less than 3 will be included in each CPT group. When the waitlist control group reaches the treatment phase, if the participant count fall below 3, additional participants will be enrolled to maintain sufficient numbers. Data collection during treatment will mirror that of the active waitlist control group. Participants will be notified via institutional mail which group they have been enrolled in.

In addition to the treatment groups, CPT and control group members will complete a PCL-5 at the beginning of each session. As well as, pre-treatment testing session two weeks prior to the start of treatment. After treatment session 5, CPT and control group members will complete mid-treatment testing assessments. Participants will be called down individually to complete these assessments in a private room with a research assistant after completing the 5th therapy session, but before completing the 8th therapy session. CPT and control group members will then complete post-treatment testing within one week after completing week 6 of treatment. One month after the treatment is completed, CPT and control group members will complete follow-up testing and interviewing about their experience in the treatment groups and will have one follow up CPT session 6-8 weeks post-treatment. Post-treatment and one-month follow up-testing will follow the same procedure as pre-treatment and mid-treatment testing. Final follow-up will occur three months after the end of treatment. Procedures will be the same as other timepoint follow-ups. CPT and control group members will be asked to complete 18 sessions in total (pre-treatment, mid- treatment, post- treatment, one-month follow up-testing, three-month follow-up treatment, 12 group sessions and one follow-up CPT session).

ELIGIBILITY:
Participants will be selected and screened from the Department of Corrections trauma treatment waitlist.

Inclusion Criteria:

* 18 years old or older
* meet PCL-5 criteria for current PTSD diagnosis within 2 months of enrollment
* no scheduled release date before the end of the treatment group
* able to understand the consent form as measured by the consent quiz
* have not participated in the previous CPT groups with UW project
* No active symptoms of psychosis that would interfere with the individual's ability to participate in the group
* No active suicidal ideation with intent or plan
* Able and willing to participate in group therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD Checklist for DSM-5 (PCL-5) severity score | baseline (two weeks prior to intervention), up to 6 weeks (mid-intervention), up to 13 weeks (one week post-intervention), up to 18 weeks (one month post-treatment), and up to 26 weeks (three months post-treatment)
  PTSD symptom severity is measured by PCL-5 questionnaire (scores from 0, no symptoms, to 80, high severity); primary measure of intervention efficacy

SECONDARY OUTCOMES:
Change in score on the Beck Depression Inventory 2 (BDI-II) | baseline (two weeks prior to intervention), up to 6 weeks (mid-intervention), up to 13 weeks (one week post-intervention), up to 18 weeks (one month post-treatment), and up to 26 weeks (three months post-treatment)
  Depression level measured by score on BDI-II (between 0 and 63; over 40 = extreme depression); secondary measure of intervention efficacy
Change in score on the Beck Anxiety Inventory (BAI) | baseline (two weeks prior to intervention), up to 6 weeks (mid-intervention), up to 13 weeks (one week post-intervention), up to 18 weeks (one month post-treatment), and up to 26 weeks (three months post-treatment)
  Anxiety level measured by score on BAI (between 0 and 63; over 30 = severe anxiety); secondary measure of intervention efficacy
Percentage of participants endorsing 2 or higher on Q9 of BDI-II | baseline (two weeks prior to intervention), up to 6 weeks (mid-intervention), up to 13 weeks (one week post-intervention), up to 18 weeks (one month post-treatment), and up to 26 weeks (three months post-treatment)
  Question 9 on the BDI-II assesses for suicidal ideation. A score of 2 (I would like to kill myself) or 3 (I would kill myself if I had the chance; the highest score) indicate heightened levels of suicidal ideation. Participants who endorse current suicidal ideation will be referred to mental health services within the institution.
Ratings from 0-5 by clinical supervisors on therapist adherence to five session elements | Up to 7 weeks (by the end of the 12th session)
  Higher ratings indicate better adherence to session elements. Assesses for therapist adherence to CPT guidelines as secondary measure of intervention efficacy. For each 12-session intervention, 2 sessions will be audiotaped and rated.
Ratings 1-7 by clinical supervisors on quality of session elements delivered by therapist | Up to 7 weeks (by the end of the 12th session)
  Higher ratings indicate higher-quality session element (scores 1-7;1="not satisfactory", 4="satisfactory", 7="excellent") by the clinical supervisors. Competence ratings will be collected for two audiotaped group sessions out of each 12-session intervention. Assesses for therapist compliance as secondary measure of intervention efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Koenigs, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Psychiatric Institute and Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James, D.J. and L.E. Glaze, Mental health problems of prison and jail inmates, U.S.D.o. Justice, Editor. 2006: Bureau of Justice Statistics Special Report.
- [Background] Egeressy A, Butler T, Hunter M. 'Traumatisers or traumatised': Trauma experiences and personality characteristics of Australian prisoners. Int J Prison Health. 2009;5(4):212-22. doi: 10.1080/17449200903343209. PMID 25757522
- [Background] Campbell CA, Albert I, Jarrett M, Byrne M, Roberts A, Phillip P, Huddy V, Valmaggia L. Treating Multiple Incident Post-Traumatic Stress Disorder (PTSD) in an Inner City London Prison: The Need for an Evidence Base. Behav Cogn Psychother. 2016 Jan;44(1):112-7. doi: 10.1017/S135246581500003X. Epub 2015 Feb 20. PMID 25697197
- [Background] Resick, P.A., C.M. Monson, and K.M. Chard, Cognitive Processing Therapy for PTSD: A Comprehensive Manual. 2016: Guilford Press.
- [Background] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Background] Morgan RD, Winterowd CL. Interpersonal process-oriented group psychotherapy with offender populations. Int J Offender Ther Comp Criminol. 2002 Aug;46(4):466-82. doi: 10.1177/0306624X02464008. PMID 12150085